CLINICAL TRIAL: NCT00257894
Title: Baclofen Effects on Smoking Urge and Withdrawal
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment was completed with insufficient sample size for publishable results
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEUA-029-04F
Record Dates: First submitted 2005-11-21; First posted 2005-11-23 (Estimated); Results first posted 2015-11-04 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-10

CONDITIONS: Nicotine Use Disorder; Nicotine Dependence; Smoking; Tobacco Use Disorder
Keywords: Baclofen; Conditioning, Classical; Nicotine; Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Baclofen; Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baclofen condition (Experimental): Baclofen taken orally for 12 days total up to 40 mg/day maximum, divided into 3 equal portions each day. Participants receive 12 mg/day the first 3 days, 30 mg/day the next 3 days, and 40 mg/day on Days 7, 8, 9. Testing is on day 10 after the first dose is taken, with downward titration days 10-12 of 30 mg on Day 10, 20 mg on Day 11 and 10 mg on Day 12.
  Interventions: Drug: Baclofen
- Placebo condition (Placebo Comparator): Placebo capsules identical to active medication, 3/day for 12 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baclofen — Dosing taken orally for a total of 12 days: 40mg/day vs. 0mg/day (placebo tabs). The 40mg condition will receive 15mg/day the first 3 days(Days 1,2,3), 30mg/day for 3 days(Days 4,5,6), and 40mg/day for 3 days(Days 7,8,9). Downward titration: 40mg/day condition will receive 40mg/day(Day 10), 20mg/day(Day 11), and 10mg/day(Day 12).
  Other Names: Seroquel
  Arms: Baclofen condition
Drug: Placebo — Matched placebo capsules containing inert filler taken orally for a total of 12 days
  Arms: Placebo condition

SUMMARY:
The purpose of this study is to determine whether baclofen is effective in reducing smoking urge, withdrawal, and reinforcement in moderate to heavy cigarette smokers.

DETAILED DESCRIPTION:
OBJECTIVES: The long-term objective of this research program is to improve treatments for tobacco smokers by investigating the effects of medications on self-reported and psychophysiological responses to smoking cues and on behavioral-economic measures of smoking reinforcement during a period of tobacco deprivation. The specific objectives of the present application are to investigate the dose-response effects of baclofen (a gamma-aminobutyric acid B agonist), 1) on urge, and withdrawal, and 2) on the reinforcement value of smoking as measured by choices for puffs on cigarettes versus an alternative reinforcer among current smokers after 4 hours of smoking deprivation. RESEARCH PLAN: The study will use a randomized placebo-controlled between-subjects design with 64 smokers to investigate the effects of placebo and two doses (20 or 40 mg/day) of baclofen on urge to smoke and withdrawal and on choices for smoking versus money after 4 hours of deprivation. METHODS: Participants will be healthy people who smoke at least 10 cigarettes per day and who are motivated for future smoking cessation. On Day 0, a baseline session will occur after 4 hours of smoking deprivation and on Day 10 of medication the same assessments will be repeated after the final medication dose has been stabilized for at least 3 days and after 4 hours of supervised smoking deprivation has occurred. Medication differences in urge and withdrawal and in the reinforcement value of smoking cigarettes will be investigated. Dependent measures of urge and withdrawal will be by self-report. The dependent measure of reinforcement value is the ratio of choices for cigarette puffs versus money during a subsequent 2-1/2 hr period. The choice procedure will clarify the relative reinforcement value of smoking while controlling for non-specific decreases in general activity level resulting from sedation. Nicotine self-administration during the medication period will be quantified using saliva cotinine, as a secondary effect. CLINICAL RELEVANCE: More effective interventions for tobacco use could result in less suffering and mortality and in considerable savings in health care costs associated with cardiovascular disease, pulmonary disorders, and cancer.

ELIGIBILITY:
Inclusion Criteria:

* Smoke at least 10 cigarettes per day for at least 6 months and considering quitting smoking in the next 6 months-

Exclusion Criteria:

* Planning to attempt smoking cessation within the next 4 months
* Weight less than 110 lbs. or above 220 lbs.
* Use of tobacco products other than cigarettes in the previous month.
* History of: Kidney disease, uncontrolled conditions (e.g., cardiac disease, pulmonary disease, diabetes, hypertension) Neurological disease (including stroke, mini-stroke, brain injury, Alzheimers Disease, encephalitis, meningitis, seizure disorder),Phenylketonuria Schizophrenia, Schizoaffective Disorder, Paranoid Disorder, or Schizotypal Disorder.
* Current alcohol and/or drug use disorder as indicated by a screening questionnaire, past treatment for alcohol or substance use problems unless in remission(clean and sober for past year or more) or intention to seek treatment in the next 6 months for alcohol or substance use problems.
* For women: Pregnancy, nursing, not using a reliable form of birth control.
* Allergy to baclofen, Lioresal, or Kemstro.
* Taking the following medications: antidepressants(excluding selective serotonin reuptake inhibitors), bupropion, phenothiazines, antihistamines, sedative/hypnotics, benzodiazepines, alpha blockers, beta blockers.
* Lives with someone enrolled in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2005-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Damaris Rohsenow, PhD, Principal Investigator — VA Medical Center, Providence
Locations (1):
- VA Medical Center, Providence, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were veterans recruited from the Veterans Affairs Medical Center, Veterans Affairs Medical Center staff, visitors, and smokers recruited from the community.
Pre-assignment Details: Nine people washed out or failed to return before assignment to groups, or were assessed with an invalid informed consent so the IRB required their data to be excluded from all analyses, and no demographic information is available on these people, leaving n = 32 with at least age and gender.
Period: Overall Study
Arm/Group | Baclofen Condition | Placebo Condition
Started | 21 | 20
Completed | 17 | 15
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baclofen Condition | Placebo Condition | Total
Number analyzed (Participants) | 17 | 15 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (10.7) | 43.5 (9.8) | 45.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 11 | 8 | 19
Region of Enrollment [Number; unit: participants]
  United States | 17 | 15 | 32
Fagerstrom Test for Nicotine Dependence [Mean (Standard Deviation); unit: units on a scale] — The total score of a measure of behaviors indicating tobacco dependence, with a range from 0 (least dependent) to 10 (most dependent).
  units on a scale | 6.18 (1.59) | 5.93 (2.76) | 6.06 (2.18)
Number of cigarettes smoked per day [Mean (Standard Deviation); unit: cigarettes] | 20.4 (7.6) | 19.0 (8.1) | 19.7 (7.8)
Number of years smoked daily [Mean (Standard Deviation); unit: years] | 28.5 (11.9) | 24.9 (11.7) | 26.9 (11.7)

OUTCOME MEASURES:

1. Primary Outcome: Total Score on Questionnaire of Smoking Urges
Description: Questionnaire of Smoking Urges assesses cravings to smoke. the score is the mean of 10 7-point Likert ratings so the range of the total score is from 1 (no urge) to 7 (intense urge).
  These data are only available on the subset of participants who participated through Day 10.
Time Frame: Measures are assessed on the tenth day of medication titration, after 5 hours of smoking deprivation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baclofen Condition | Placebo Condition
Number analyzed (Participants) | 16 | 11
units on a scale | 5.5 (2.1) | 5.3 (2.3)
Statistical Analysis 1: Comparison: Baclofen Condition vs Placebo Condition; Test type: Superiority or Other; p = .57, ANOVA — Effect size close to zero (eta squared of .01); Interaction effect term from group by time ANOVA

2. Secondary Outcome: Nicotine Self-administration as Quantified by Carbon Monoxide Boost During a Behavioral Self-administration Task.
Description: Expired carbon monoxide (CO) assessed before and after a 2.5-h period when they make choices for cigarette puffs versus money. CO Boost is the difference score, possibly ranging from -25 (improved) to +25 (worse).
  These data are only available on the subset of participants who participated through Day 10..
Time Frame: Measures are assessed on the tenth day of medication titration, after 5 hours of smoking deprivation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baclofen Condition | Placebo Condition
Number analyzed (Participants) | 16 | 11
units on a scale | 4.69 (4.16) | 5.27 (5.90)
Statistical Analysis 1: Comparison: Baclofen Condition vs Placebo Condition; Test type: Superiority or Other; p = .60, ANOVA — Effect size about zero (eta squared = .01); Interaction term from a group by time ANOVA

3. Secondary Outcome: Cigarette Choice Task
Description: At 20 times spaced over a 2.5 h period, participants chose between smoking two puffs (of pre-determined size) of a cigarette and receiving US$0.10. The primary behavioral outcome measure was number of cigarette choices, ranging from 0 (no smoking) to 20 (smoking the most allowed).
  These data are only available on the subset of participants who participated through Day 10.
Time Frame: Tenth day of medication titration
Measure: Mean (Standard Deviation); unit: choices
Arm/Group | Baclofen Condition | Placebo Condition
Number analyzed (Participants) | 16 | 11
choices | 15.4 (5.7) | 18.2 (4.8)
Statistical Analysis 1: Comparison: Baclofen Condition vs Placebo Condition; Test type: Superiority or Other; p = .79, ANOVA — Effect size (eta squared) = 0; Interaction term of a group by time ANOVA

4. Primary Outcome: Minnesota Nicotine Withdrawal Questionnaire
Description: Measure of degree of nicotine withdrawal at the time. Scored as the mean of 8 5-point ratings so the total score ranges from 0 (no withdrawal) to 4 (severe withdrawal).
  These data are only available on the subset of participants who participated through Day 10.
Time Frame: Day 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baclofen Condition | Placebo Condition
Number analyzed (Participants) | 16 | 12
units on a scale | 1.06 (1.73) | 1.58 (2.35)
Statistical Analysis 1: Comparison: Baclofen Condition vs Placebo Condition; Analysis of variance, group by time (Day 0 vs. Day 10); Test type: Superiority or Other; p = .21, ANOVA — For test of drug by time interaction effect; Medium effect size, eta squared = .061

ADVERSE EVENTS:
Time Frame: 1 year 11 months
Description: Jan. 2007 - Nov. 2008
Arm/Group | Baclofen Condition | Placebo Condition
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baclofen Condition (N=21) | Placebo Condition (N=20)
Hospitalization (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Broke wrist when in a domestic altercation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No